CLINICAL TRIAL: NCT03146377
Title: An Open-label, Single-centre, Single-arm Phase II Study of Triplet Combination of Capecitabine, Oxaliplatin and Irinotecan (Xeloxiri) as Salvage Therapy in Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Study of Xeloxiri Regimen for Patients With Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. YAU Chung Cheung Thomas, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MONC-LGI05
Record Dates: First submitted 2014-05-06; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xeloxiri (Experimental)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Capecitabine — 1250 mg/m2 BD orally for 1 week of a 2-week cycle (i.e. 1 week on, 1 week off)
  Other Names: Xeloda
Drug: Oxaliplatin — 85 mg/m2 IV on day 1 of a 2-week cycle
Drug: Irinotecan — 165 mg/m2 IV on day 1 of a 2-week cycle

SUMMARY:
This is an open-label, single centre, single-arm phase II study which aims to assess the efficacy and tolerability of triplet combination of capecitabine, oxaliplatin and irinotecan (Xeloxiri regimen) in treating patients with refractory metastatic colorectal cancer. Clinical data from patients diagnosed with colorectal cancer will be collected and analyzed in this study. The patients' data will be collected and maintained in the Division of medical oncology of the Department of Medicine, Queen Mary Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age, male or female.
* Histopathologically or cytologically confirmed adenocarcinoma.
* Failed ≥ 2 lines of standard therapy which must include a fluoropyrimidine, oxaliplatin and/or irinotecan, administered either as monotherapy or doublets.
* ECOG performance status 0 to 2.
* Adequate bone marrow reserve.
* Absolute neutrophil count > 1 × 109/L.
* Total bilirubin < 3 × the upper limit of the normal range.
* Life expectancy ≥ 12 weeks.
* Signed written informed consent form.

Exclusion Criteria:

* Prior malignant disease other than colorectal cancer within 5 years of study entry.
* Patients suitable for surgical or locoregional therapies.
* Patients unable to swallow oral medications.
* Any evidence of brain metastasis (unless the patient is >6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry).
* Active clinically serious infections (> grade 2 NCI / CTC Adverse Event version 3.0).
* History of allergy to platinum compounds.
* Patients who have chronic inflammatory bowel disease and/or bowel obstruction.
* Patients who have severe bone marrow failure.
* Patients undergoing renal dialysis.
* History of HIV infection.
* Seizure disorder requiring medication (such as steroids or anti-epileptics).
* Women who are pregnant or breast-feeding, or women of child-bearing potential who are unable or unwilling to practice a highly effective means of contraception.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Change from baseline in size approximately every 8 weeks (4 cycles), up to approximately 12 months

SECONDARY OUTCOMES:
Progression-free survival | From date of start until the date of first documented progression or death from disease-related causes or last follow-up, whichever came first, assessed up to 18 months
Overall survival | From date of start until the date of death from any cause or last follow-up, whichever came first, assessed up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yau, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong